CLINICAL TRIAL: NCT03042403
Title: Effects of the Breath Stacking Technic in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Luciene Aparecida José Vaz, physiotherapist, Federal University of Uberlandia
Other Study IDs: CEP/UFU 364/11
Record Dates: First submitted 2017-01-24; First posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Hemodynamic Instability
Keywords: hemodynamics; physiotherapy; breath stacking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breath stacking: During initial rest period, the volunteer remained seated for 10' in spontaneous breathing. During carrying out of the breath stacking technic, the volunteer remained seated, being requested to hold the mask on his/her face not allowing air scape, The volunteer was oriented to inhale normally and exhale all the air during expiration for 20 seconds. During the 20 seconds of applying of technic, in the three series the maximum inspiratory and expiratory pressures reached during the carrying out of technic. In the final rest period, right after technic end, the volunteers remained seated for 10 minutes in spontaneous breathing and again the same variables of control at the 10th minute were assessed.
  Interventions: Other: Breath stacking

INTERVENTIONS:
Other: Breath stacking — During initial rest period, the volunteer remained seated for 10' in spontaneous breathing. Right after, the measurement of arterial pressure, of SpO2 (%), of heart rate, of respiratory frequency and applied to a modified effort perception Borg. During carrying out of the breath stacking technic, the volunteer remained seated, being requested to hold the mask on his/her face not allowing air scape, The volunteer was oriented to inhale normally and exhale all the air during expiration for 20 seconds, and the variables were assessement again the same variables of control. In the final rest period, right after technic end, the volunteers remained seated for 10 minutes in spontaneous breathing and again the same variables of control at the 10th minute were assessed.

SUMMARY:
This study aims to Analyze and compere the hemodynamic and respiratory variables before, during and after the applying of technic as well as evaluate respiratory pressures generated during applying of this same technic and correlate them with the effort noticed by device user.

DETAILED DESCRIPTION:
The breath stacking technic (BS) is an inspiratory maneuver used for recruitment of collapsed alveoli and, consequently, improves oxygenation and, therefore, used by respiratory physiotherapy aiming promoting lung re-expansion being. The BS was described by Marini as an attempt of optimizing vital capacity in little co-operative individuals and hemodynamics has been considered a way of incentive spirometry that provides high lung volume, in situations, in which, inspiratory maneuver duration can be as important as the volume reached, composing an alternative incentive of inspiration technic4. The system used is composed by an interface (facial mask) connected to the patient, an inspiratory unidirectional valve and the respiratory branch which is kept occluded during the carrying out of maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 to 30, sedentary, absence of neuromuscular and/or cardiac respiratory diseases

Exclusion Criteria:

* the smokers, overweight, claustrophobic or the ones with difficulty in carrying out the technic

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 52 healthy young volunteers The volunteers at the age of 18 to 30, sedentary: absence of neuromuscular and/or cardiac respiratory diseases were included, the smokers, overweight, claustrophobic or the ones with difficulty in carrying out the technic were excluded
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
maximum inspiratory and expiratory pressures | During the intervention. They will be used to verify the average pressures generated during the execution of the technique. Time of the technique equal to 20 seconds.
  connected to a manometer from brand Commercial Medica (Brazil) used to measure maximum inspiratory and expiratory pressures generated during carrying out of technic. The volunteer was oriented to inhale normally and exhale all the air during expiration for 20 seconds.

SECONDARY OUTCOMES:
modified effort perception Borg scale | Before, during and after the intervention. They will be used to compare the variation before, during and after the technique. Valuation time was 1 minute.
  applied to a modified effort perception Borg scale with a score from 0 to 10, considering 0 the smallest effort noticed and 10 the biggest effort reported
heart rate | Before, during and after the intervention. They will be used to compare the variation before, during and after the technique. Valuation time was 1 minute.
  by palpation method of radial artery, of respiratory frequency by direct counting of thoracic movement
peripheral oxygen saturation | Before, during and after the intervention. They will be used to compare the variation before, during and after the technique. Valuation time was 1 minute.
  through a pulse oximeter
systolic arterial pressure | Before, during and after the intervention. They will be used to compare the variation before, during and after the technique. Valuation time was 1 minute.
  the measurement of systolic arterial pressure were assessed using an aneroid-type sphygmomanometer
diastolic arterial pressure | Before, during and after the intervention. They will be used to compare the variation before, during and after the technique. Valuation time was 1 minute.
  the measurement of systolic arterial pressure were assessed using an aneroid-type sphygmomanometer from the brand Lamedial Commercial

CONTACTS AND LOCATIONS:
Overall Officials: Celia R Lopes, Principal Investigator — Federal University of Uberlandia

IPD SHARING:
Plan to Share IPD: No